CLINICAL TRIAL: NCT05292885
Title: Mp-MRI in the Diagnosis of Liver Fibrosis After Liver Transplantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Other Study IDs: QYFYWZLL26786
Record Dates: First submitted 2022-03-15; First posted 2022-03-23 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Liver Fibrosis After Liver Transplantation; Multiparameter Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Gadopentetate Dimeglumine Injection — Patients with liver fibrosis after liver transplantation receive multi-parameter magnetic resonance scanning, percutaneous liver biopsy (or FibroScan).

SUMMARY:
It is an open label observation clinical trial, all participants are liver transplant patients. The investigators deem to make a better criteria for assessing liver fibrosis after liver transplantation. The point of the clinical trial is to evaluate the efficacy of multiparameter MRI in the diagnosis of liver fibrosis after liver transplantation.

DETAILED DESCRIPTION:
We collected patients aged 18 to 85 who had undergone liver transplantation. At the same time, all patients underwent liver biopsy or ultrasonic transient elastography after MRI. People who were allergic to gadolinium contrast agent, serious cardiopulmonary disease and contraindications to MRI were excluded.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 -85 years
* Patients after liver transplantation
* Patients who are going to undergo liver biopsy or ultrasonic transient elastography
* Patients voluntarily joined the study and signed informed consent

Exclusion Criteria:

* Patients with tumor
* Patients who are allergic to gadolinium contrast agent
* Patients with contraindications to magnetic resonance imaging
* Patients with severe heart and lung diseases
* Patients who are not suitable for this study according to the researcher's judgment.

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with liver fibrosis after liver transplantation underwent percutaneous liver biopsy or FibroScan.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-03-18 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Mp-MRI in the Diagnosis of Liver Fibrosis After Liver Transplantation | 03.18.2022 to12.01.2022
  Mp-MRI as a PET-CT biomarker to Liver Fibrosis after Liver Transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Guangjie Yang, PhD, Study Chair — The affiliated hostpital of Qingdao University
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China